CLINICAL TRIAL: NCT00921258
Title: Active Control of Prostatic Cancer With Criteria of Latence. Impact on Specific 10 Years Survival.
Brief Title: Active Control of Prostatic Cancer With Criteria of Latence
Acronym: SURACAP
Status: Terminated | Type: Observational
Why Stopped: Financial problem (not enough budget to continue the study)
Sponsor: Clinique Mutualiste Chirurgicale de la Loire (Other)
Responsible Party: Sponsor
Other Study IDs: 0700043; 2007-A00871-52
Record Dates: First submitted 2009-06-12; First posted 2009-06-16 (Estimated); Last update posted 2015-06-04 (Estimated); Status verified 2015-06

CONDITIONS: Prostate Cancer
Keywords: latent prostate cancer; Patient with latent prostate cancer; PSA ≤ 10 ng/ml; Clinical stage T1c or T2a; Patient who accept just be control
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- control group: Patient with latent prostate cancer who agree to be controled instead of to be treated
  Interventions: Procedure: prostate biopsy

INTERVENTIONS:
Procedure: prostate biopsy — patient of control group will have :
  * 1 prostate biopsy 3 months after diagnostic biopsy
  * 1 prostate biopsy each year during 2 years
  * 1 prostate biopsy each 2 years during 8 years

SUMMARY:
This study concern a prospective cohort pf patients with latent prostate cancer. We study the specific survival at 10 years of patients who accept an active control.Patients inclusion are realized in 2 stages:

* patient with inclusion criteria (PSA < 10 ng/ml, clinical stage T1c or T2a, Gleason < or = 6) are registered if they accept a second prostate biopsy in a 3 months delay
* after analyse of second biopsy in central laboratory and confirmation of latent prostate biopsy, patients are included if they accept active control Included patients will have 1 biopsy by years the first two years and then 1 biopsy each 2 years during 8 years.

If progression of cancer happens during the 10 years control, active control will be stopped and patient will be treated by surgery and chemotherapy.

DETAILED DESCRIPTION:
This study concern the active control during 10 years of patient with latent prostate cancer who accept not be treated immediately.

ELIGIBILITY:
Inclusion Criteria:

* patient with a latent prostatic cancer
* aged less 75 years old,
* life expectation higher than 10 years
* Clinic statue T1c or T2a
* with a seric PSA (prostatic specific antigen)smaller than 10ng/ml
* more than 10 biopsy cores samples
* patient with less than 3 cores samples with tumor and none care sample with more than 3mm of tumor
* Gleason score inferior at 7
* patient's agreement about project and a second biopsy which will include definitive patient: realized 3 months after the first and having: 14 biopsy cores samples (10 like previously and 4 more specific: taking around the positives initials biopsies), less than 3 cores samples with tumor, ,any cores samples with more than 3mm of tumor, a Gleason score superior at 7.

Exclusion Criteria:

* patient aged 75 years old and more
* no patient's agreement
* lack of understanding of plan
* patient with guardianship
* life expectation smaller than 10 years
* patient with an other cancer less than 5 years
* Local clinical statue greater than T2a
* seric PSA higher than 10ng/ml
* less than 10 biopsies
* more than 2 positives biopsies during the first intervention
* 3 cores samples with more than 3mm of tumor
* 4th grade on the biopsies
* patient's refuse to realize the second biopsies
* patient who ask a treatment after the first medical examination
* patient with less 4 special biopsies around the previously initial cores samples or more than 2 positives biopsies or biopsies with more than 3mm of tumor or patient having a 4 grade on biopsies, during the second medical examination.

Ages: 18 Years to 74 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with latent prostate cancer who agree to be controlled instead of to be immediately treated for this cancer
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2007-12; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Evaluates specific survival to 10 years | 10 years

SECONDARY OUTCOMES:
To evaluate acceptation of 2nd biopsy to confirm latent cancer | 10 years
To evaluate global survival of patient in control | 10 years
To evaluate the survival of patient with a secondary active treatment after a control period | 10 years
To evaluate delay to secondary treatment after a period control | 10 years
To evaluate survival rate without biological or clinical progression of cancer | 10 years
To evaluate quality of life | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas MOTTET, Dr, Principal Investigator — Clinique Mutualiste Chirurgicale
Locations (15):
- France (15):
  - R Azzouzi, Angers
  - Jean-Louis DAVIN, Avignon
  - Henri BENSADOUN, Caen
  - SALOMON, Créteil
  - René GASCHIGNARD, La Roche-sur-Yon
  - RUFFION, Lyon
  - Eric LECHEVALLIER, Marseille
  - P. ROSSI, Marseille
  - Xavier REBILLARD, Montpellier
  - RIGAUD Jérôme, Nantes
  - Christophe AVANCES, Nîmes
  - IRANI Jacques, Poitiers
  - P Colloby, Pontoise
  - Clinique Mutualiste Chirurgicale, Saint-Etienne
  - SOULIE Michel, Toulouse